CLINICAL TRIAL: NCT02077556
Title: The Effect of Everolimus on the Pharmacokinetics of Tacrolimus in Renal Transplant Patients, and the Effect of ABCB1、CYP3A4、CYP3A5、PORGenetic Polymorphism on the Two Drugs
Brief Title: Effect of Everolimus on the Pharmacokinetics of Tacrolimus in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201312011MINA
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2018-07

CONDITIONS: Drug Interaction Potentiation
Keywords: tacrolimus, everolimus, pharmacokinetics, drug interaction
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Tacrolimus; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Experimental): Everolimus/Tacrolimus/Methylprednisolone & Prednisolone
  Interventions: Drug: Everolimus; Drug: Tacrolimus; Drug: Methylprednisolone; Drug: Prednisolone
- Mycophenolate mofetil (Active Comparator): Mycophenolate mofetil/Tacrolimus/ Methylprednisolone & Prednisolone
  Interventions: Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Methylprednisolone; Drug: Prednisolone

INTERVENTIONS:
Drug: Everolimus — Everolimus: 1 mg orally every 12 hours from post-operation day 1 to achieve trough concentrations of 3-8 ng/mL
  Other Names: Certican
  Arms: Everolimus
Drug: Mycophenolate mofetil — Mycophenolate mofetil: 10-15 mg/kg orally every 12 hours from post-operation day 1 (decrease 50% dose if white blood cell < 4000/mcL)
  Other Names: CellCept
  Arms: Mycophenolate mofetil
Drug: Tacrolimus — Tacrolimus: 0.05-0.075 mg/kg orally every 12 hours from post-operation day 1 to achieve trough concentrations of 8-12 ng/mL
  Other Names: Prograf
Drug: Methylprednisolone — Methylprednisolone: 50 mg iv every 6 hours on post-operation day 1, 40 mg iv every 6 hours on post-operation day 2, 30 mg iv every 6 hours on post-operation day 3, 20 mg iv every 6 hours on post-operation day 4, 20 mg iv every 8 hours on post-operation day 5, 20 mg iv every 12 hours on post-operation day 6, 20 mg iv on post-operation day 7
  Other Names: Solu-Medrol
Drug: Prednisolone — Prednisolone: 20 mg orally once a day from post-operation day 8 to post-operation week 4, then titrated gradually
  Other Names: Predonine

SUMMARY:
The purpose of this study is to understand the effects of everolimus on tacrolimus pharmacokinetics (pk) in patients receiving de novo kidney transplants.

DETAILED DESCRIPTION:
Multidrug immunosuppression regimens have synergistic effects which allow the use of lower doses of individual agents. These regimens generally include calcineurin inhibitors (CNIs: cyclosporine or tacrolimus), mammalian target of rapamycin (mTOR) inhibitors (everolimus or sirolimus), and corticosteroids. CNIs and mTOR inhibitors are substrates for cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp); in addition, cyclosporine is a inhibitor of CYP3A4 and P-gp. Therefore, concomitant administration of those drugs may alter their serum levels.

It is remained to be evaluated whether the pharmacokinetics or clinical efficacy of tacrolimus will be affected when the regimens contain everolimus in clinical practice and the effect of ABCB1、CYP3A4、CYP3A5、POR genetic polymorphism on the two Drugs. Mycophenolate mofetil (MMF) has no effect on pharmacokinetics of tacrolimus; therefore, MMF is used as a control to understand the effects of everolimus on pharmacokinetics of tacrolimus in patients receiving de novo kidney transplants. The effect of ABCB1、CYP3A4、CYP3A5、POR genetic polymorphism on the two Drugs was also assessed.

ELIGIBILITY:
Inclusion criteria:

* De novo kidney transplants
* 20 - 65 years old
* aspartate aminotransferase/alanine aminotransferase within 2 times the upper limit of normal range

Exclusion criteria:

* Pregnancy
* Tuberculosis
* Hepatitis B or C carrier status
* Human immunodeficiency virus-positive status
* Retransplantation or multiorgan transplantation
* History of rheumatoid arthritis
* Use of drugs that might have enhanced or inhibited CYP3A4 or P-gp activity

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profiles | Post-operation day 8-10
  Pharmacokinetic parameters include the maximum concentration, trough concentration, area under the whole-blood concentration-time curve between 0 and 12 hours, time to maximum concentration, volume of distribution at steady state, and clearance at steady state.

SECONDARY OUTCOMES:
Acute rejection | Within the first 2 weeks post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Kun Tsai, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan